CLINICAL TRIAL: NCT02164981
Title: A Randomized Double-Blind, Placebo-Controlled, Proof of Concept Study of Intravenous Sodium Nitroprusside in Adults With Symptomatic Schizophrenia
Brief Title: A Proof of Concept Study of Intravenous Sodium Nitroprusside in Adults With Symptomatic Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Director, Clinical Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014P001204; NCT02695589 (obsolete NCT alias)
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Nitroprusside; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Drug - Drug (Active Comparator): Phase 1 - intravenous sodium nitroprusside Phase 2 - intravenous sodium nitroprusside
  Interventions: Drug: sodium nitroprusside
- Placebo - Drug (Other): Phase 1 - intravenous dextrose Phase 2 - intravenous sodium nitroprusside
  Interventions: Drug: sodium nitroprusside
- Placebo - Placebo (Placebo Comparator): Phase 1 - intravenous dextrose Phase 2 - intravenous dextrose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: sodium nitroprusside — intravenous
  Other Names: Nitropress
  Arms: Drug - Drug; Placebo - Drug
Other: Placebo — Placebo
  Other Names: 5% dextrose
  Arms: Placebo - Placebo

SUMMARY:
The primary objective of this study is to investigate whether a single infusion of intravenous sodium nitroprusside (0.5 μg/kg/min for 4 hours) is superior to placebo (5% dextrose solution) at in treating positive and negative symptoms of schizophrenia

DETAILED DESCRIPTION:
This is a phase II proof of concept (POC), multi-center, prospective, randomized, placebo-controlled, Sequential Parallel Comparison Design (SPCD) study, in which a total of 60 subjects with schizophrenia will be enrolled.

The study will be conducted in two stages. The study treatment will be administered in a double-blind fashion for all subjects throughout both stages of the study. A total of 60 subjects with schizophrenia will be randomized in a 1:1:1 ratio to drug-drug sequence [n=20; i.v. sodium nitroprusside (0.5 μg/kg/min for 4 hours) at week 0 and week 2], placebo-drug sequence [n=20; i.v. placebo at week 0 and i.v. sodium nitroprusside (0.5 μg/kg/min for 4 hours) at week 2], and placebo-placebo sequence [n=20; i.v. placebo at week 0 and again at week 2]. The 4-week double-blind phase of treatment will be divided into two phases: Phase 1, from week 0 to week 2, and Phase 2 from week 2 to week 4. At the end of Phase 1 (week 2), the randomized subjects will be assessed and categorized into responders and non-responders, based on 20% or more reduction from baseline in their PANSS total score as per the evaluations at Randomization Visit (week 0). The data from the patients deemed placebo non-responders in phase 1 who go on to either stay on placebo or to receive treatment with sodium nitroprusside will be pooled with the data from Phase 1 from all subjects, according to SPCD.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be eligible for this study:

1. Males or Females aged 18-65 years inclusive.
2. Primary diagnosis of Schizophrenia established by a structured psychiatric evaluation (SCID) based on Diagnostic and Statistical Manual of Mental Disorders Forth Edition (DSM-IV-TR) criteria.
3. Written informed consent in compliance with 21 CFR part 50 and in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guidelines.
4. A Positive and Negative Syndrome Scale (PANSS) (Kay et al., 1994) total score ≥ 70 with a score of > 4 on two or more of the following PANSS items: delusions, conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content.
5. A score of ≥4 on the Clinical Global Impression-Severity (CGI-S) (Guy, 1976).
6. Confirmation of both diagnosis and severity of psychosis symptoms by an independent MGH SAFER interview.
7. Must have ongoing antipsychotic treatment for at least 8 weeks, with a stable dose for at least 4 weeks. Subjects who have failed to achieve clinically-recognized symptom reduction to at least 1 marketed antipsychotic agent, given at a Physician Desk Reference (PDR)-defined therapeutic dose for ≥ 8 weeks during the past 12 months, as assessed by the MGH FAST, will be eligible
8. Understands and is able, willing, and (in the opinion of the investigator) likely to fully comply with the study procedures and restrictions.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from the study:

1. Subjects with a history of renal insufficiency, congestive heart failure, cardiac arrhythmias or history of myocardial infarction.
2. Subjects with a history of symptomatic orthostatic hypotension defined as sitting to standing systolic blood pressure < 90mmHg or diastolic blood pressure < 60mm Hg with any of the following symptoms: lightheaded or dizzy upon standing, blurry vision, weakness, fainting (syncope), confusion, or nausea.
3. Subjects with any clinically significant abnormalities as determined by medical history, physical exam, clinical and lab evaluation suggestive of an underlying disease state that may, in the opinion of the investigator, confound the results of study, increase risk to the subject, or lead to difficulty complying with the protocol.
4. Subjects on chlorpromazine, PDE-5 inhibitors, nitrites and any medication with CNS effects with the exception of antipsychotic drugs (other than chlorpromazine) anticholinergics, b-adrenergic antagonists, amantadine, biperiden, diphenhydramine, lorazepam, zolpidem, and temazepam.
5. Medications which in the opinion of the PI, and in conjunction with the medical monitor, may be expected to significantly interfere with the metabolism or excretion of sodium nitroprusside, and/or may be associated with a significant drug interaction with sodium nitroprusside that may pose a significant risk to subjects' health and/or confound the study data.
6. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed at screening visit prior to randomization and prior to baseline at visits 3 and 6. Women enrolled in this trial must use adequate birth control.
7. Subjects with a current (within the last 3 months) DSM-IV-TR diagnosis of alcohol or substance use disorder or dependence (excluding nicotine) as established by the clinical assessment (SCID) at the screening visit will be excluded.
8. Has tested positive for any of the following: cannabis, opioids, cocaine, amphetamines, barbiturates methadone, methamphetamine and phencyclidine at the screening or baseline visits. If positive, the urine drug toxicology screen may be repeated once based on investigator judgment, but due to safety concerns, the result must be negative for the subject to continue in the study.
9. Subjects at imminent risk of suicide or injury to self or others, as per the opinion of the investigator, or history of significant suicide attempt within the last 6 months as per C-SSRS.
10. Subjects that have taken an investigational drug or taken part in a clinical trial within 30 days prior to screening.
11. Any other reason that, in the opinion of the investigator, would compromise patient safety or integrity of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05-01; Primary Completion 2017-03-31 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital; Roy Perlis, MD MSc, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Schizophrenia Clinical Research Program, Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Zucker Hillside Hospital, Glen Oaks, New York
  - New York University Langone Medical Center/Bellevue Hospital, New York, New York

REFERENCES:
- [Derived] Brown HE, Freudenreich O, Fan X, Heard SO, Goff D, Petrides G, Harrington AL, Kane JM, Judge H, Hoeppner B, Fava M, Perlis RH. Efficacy and Tolerability of Adjunctive Intravenous Sodium Nitroprusside Treatment for Outpatients With Schizophrenia: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Jul 1;76(7):691-699. doi: 10.1001/jamapsychiatry.2019.0151. PMID 30916714

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per the Sequential Parallel Comparison Design, the 18 subjects in the SNP-SNP group were excluded from Phase 2 analyses. There were no Phase 1 placebo responders, so no exclusions were made based on this SPCD criterion. Ph 1 (N=52): all groups; Ph 2 (N=34): (Placebo)-Placebo (N=18), (SNP)-Placebo (N=16). All subjects were followed for 28 days.
Groups:
- Drug - Drug: Phase 1 - intravenous sodium Nitroprusside (Drug) Phase 2 - intravenous sodium Nitroprusside (Drug)
  Subjects will receive i.v. sodium nitroprusside (0.5 μg/kg/min for 4 hours) at Day 0 (Phase 1) and Day 14 (Phase 2)
- Placebo - Drug: Phase 1 - intravenous dextrose (Placebo) Phase 2 - intravenous sodium Nitroprusside (Drug)
  Subjects will receive i.v. placebo (intravenous dextrose) at Day 0 (Phase 1) and i.v. sodium nitroprusside (0.5 μg/kg/min for 4 hours) at Day 14 (Phase 2)
- Placebo - Placebo: Phase 1 - intravenous dextrose (Placebo) Phase 2 - intravenous dextrose (Placebo)
  Subjects will receive i.v. placebo (intravenous dextrose) at Day 0 (Phase 1) and again at Day 14 (Phase 2).
Period: Started
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
Started | 23 | 19 | 18
Completed (These subjects moved onto the Phase 1) | 18 | 16 | 18
Not Completed | 5 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0
Period: Phase 1 (Day 0 - Day 14)
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
Started | 18 | 16 | 18
Completed | 18 | 14 | 18
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0
Period: Phase 2 (Day 14 - Day 28)
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
Started | 18 | 14 | 18
Completed | 16 | 12 | 18
Not Completed | 2 | 2 | 0
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo | Total
Number analyzed (Participants) | 18 | 16 | 18 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (10.5) | 45.9 (12.3) | 40.4 (11.0) | 44.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 14 | 12 | 14 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 17 | 15 | 16 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 9 | 6 | 25
  Black | 6 | 5 | 11 | 22
  Asian | 1 | 2 | 1 | 4
  Other | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 16 | 18 | 52
The Positive and Negative Syndrome Scale (PANSS) at Baseline (Day 3) [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Syndrome Scale (PANSS) is a 30-item questionnaire used to evaluate schizophrenia symptoms; consisting of Positive (7 items), Negative (7 items), and General Psychopathological scales (16 items) sections. Each item (symptom) is scored on a 7-point scale, higher scores representing increasing levels of psychopathology: Positive scale: 7 Items, (min. score = 7, max. score = 49); Negative scale: 7 Items, (min. score = 7, max. score = 49). For this measure, only the positive and negative scales are included in the total score (min. total score = 14, max., score = 98)
  units on a scale
    PANSS -total | 83.6 (10.0) | 77.6 (8.8) | 81.7 (8.8) | 80.9 (9.2)
    PANSS - positive | 24.9 (3.5) | 22.3 (3.4) | 22.6 (3.1) | 23.26 (3.3)
    PANSS - negative | 20.9 (5.5) | 20.3 (5.0) | 21.4 (4.6) | 20.8 (15.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) - Total Score - Study Phases 1 and 2
Description: The Positive and Negative Syndrome Scale (PANSS) will be used to measure symptom severity in this trial. PANSS is a 30-item questionnaire used to evaluate schizophrenia symptoms, based on the clinical interview as well as reports of family members or primary care hospital workers. PANSS consists of Positive scale (7 items), Negative scale (7 items), and General Psychopathological scale (16 items) sections. Each item (symptom) will be scored on a 7-point scale with higher scores representing increasing levels of psychopathology: 1) Absent, 2) Minimal, 3) Mild, 4) Moderate, 5) Moderate severe, 6) Severe, and 7) Extreme. Total score minimum = 30, maximum = 210
Time Frame: For Phase 1, timeframe is Day 0 and Day 14; Phase 2 timeframe is Day 14 and Day 28
Population: Ph 1 analysis includes 34 subjects with Baseline PANSS data in the Placebo-Placebo (N=18) and Placebo-Drug (N=16) groups and 18 Drug-Drug group subjects. Per SPCD, the Ph 2 data excludes 18 Drug-Drug group subjects and includes the 14 subjects in the Placebo-Drug group and 18 subjects in the Placebo-Placebo group with PANSS Baseline data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Drug: Phase 1 - intravenous sodium nitroprusside Phase 2 - intravenous sodium nitroprusside
  sodium nitroprusside: intravenous
- Placebo: Phase 1 - intravenous dextrose Phase 2 - intravenous dextrose
  Placebo:
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 32 | 34
units on a scale
  Phase 1 - Total Score - Baseline: number analyzed (Participants) | 18 | 34
  Phase 1 - Total Score - Baseline | 83.6 (10.0) | 79.8 (8.9)
  Phase 1 - Total Score - Day 14: number analyzed (Participants) | 18 | 32
  Phase 1 - Total Score - Day 14 | 77.6 (12.2) | 76.7 (11.0)
  Phase 1 - Total Score - Change: number analyzed (Participants) | 18 | 32
  Phase 1 - Total Score - Change | -6.0 (11.3) | -2.5 (7.1)
  Phase 2 - Total Score - Day 14: number analyzed (Participants) | 14 | 18
  Phase 2 - Total Score - Day 14 | 74.0 (12.0) | 78.8 (10.1)
  Phase 2 - Total Score - Day 28: number analyzed (Participants) | 12 | 18
  Phase 2 - Total Score - Day 28 | 71.8 (10.6) | 74.7 (9.0)
  Phase 2 - Total Score - Change: number analyzed (Participants) | 12 | 18
  Phase 2 - Total Score - Change | -1.8 (8.2) | -4.2 (6.4)
Statistical Analysis 1: Comparison: Drug vs Placebo; Given the sequential parallel comparison design (SPCD), we used a two-stage test (weighted z-test, Tamura approach: CHANGE_score = BASELINE_value + GROUP (i.e., SNP vs. placebo)) to combine the data on treatment effects from phases 1 and 2 (weighted equally). Assessments were on Day -1 (phase 1 baseline), Day 13 (phase 1 outcome, phase 2 baseline) and Day 28 (phase 2 outcome). Only participants who at least started the infusion were included in analysis (i.e., modified intent to treat); Test type: Superiority; p = 0.57, ANCOVA — No adjustment for multiple comparisons, as there was only one primary outcome variable; Mean Difference (Final Values) = -1.04
Statistical Analysis 2: Comparison: Drug vs Placebo; The same analysis as in Analysis 1 was conducted, except that CLOZAPINE (i.e., patient used clozapine vs. other antipsychotic) was added as a covariate; Test type: Superiority; p = 0.54, ANCOVA — No adjustment for multiple comparisons, as there was only one primary outcome variable; Mean Difference (Final Values) = -1.09

2. Secondary Outcome: PANSS - Positive Subscale - Phases 1 and 2
Description: The Positive and Negative Syndrome Scale (PANSS) will be used to measure symptom severity in this trial. PANSS is a 30-item questionnaire used to evaluate schizophrenia symptoms, based on the clinical interview as well as reports of family members or primary care hospital workers. PANSS consists of Positive scale (7 items), Negative scale (7 items), and General Psychopathological scale (16 items) sections. Each item (symptom) will be scored on a 7-point scale with higher scores representing increasing levels of psychopathology: 1) Absent, 2) Minimal, 3) Mild, 4) Moderate, 5) Moderate severe, 6) Severe, and 7) Extreme. Positive scale: 7 Items, (minimum score = 7, maximum score = 49)
Time Frame: Phase 1 timeframe is Baseline and Day 14; Phase 2 timeframe is Day 14 and Day 28
Population: Ph 1 analysis includes the 34 subjects with Baseline PANSS data in the Placebo-Placebo (N=18) and Placebo-Drug (N=16) groups and 22 Drug-Drug group subjects. Per SPCD, the Ph 2 data excludes the 18 Drug-Drug group subjects and includes the 14 subjects in the Placebo-Drug group and 18 subjects in the Placebo-Placebo group with PANSS Baseline data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Drug: Phase 1 - intravenous sodium Nitroprusside or placebo Phase 2 - intravenous sodium nitroprusside
  sodium nitroprusside: intravenous
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 32 | 34
units on a scale
  Phase 1 - Positive Score - Baseline: number analyzed (Participants) | 18 | 34
  Phase 1 - Positive Score - Baseline | 24.5 (3.5) | 22.3 (3.1)
  Phase 1 - Positive Score - Day 14: number analyzed (Participants) | 18 | 32
  Phase 1 - Positive Score - Day 14 | 23.1 (4.6) | 21.3 (3.6)
  Phase 1 - Positive Score - Change: number analyzed (Participants) | 18 | 32
  Phase 1 - Positive Score - Change | -1.8 (1.8) | -0.81 (2.7)
  Phase 2 - Positive Score - Day 14: number analyzed (Participants) | 14 | 18
  Phase 2 - Positive Score - Day 14 | 20.7 (3.6) | 21.8 (3.6)
  Phase 2 - Positive Score - Day 28: number analyzed (Participants) | 12 | 18
  Phase 2 - Positive Score - Day 28 | 21.3 (4.6) | 22.3 (3.4)
  Phase 2 - Positive Score - Change: number analyzed (Participants) | 12 | 18
  Phase 2 - Positive Score - Change | 0.5 (3.8) | 0.5 (2.17)
Statistical Analysis 1: Comparison: Drug vs Placebo; Test type: Superiority; p = 0.35, ANCOVA — Exploratory efficacy outcome, hence no adjustment for multiple comparison; Mean Difference (Final Values) = -0.62
Statistical Analysis 2: Comparison: Drug vs Placebo; Test type: Superiority; p = 0.37, ANCOVA — Exploratory efficacy outcome, hence no adjustment for multiple comparisons; Mean Difference (Final Values) = -0.62

3. Secondary Outcome: PANSS - Negative Subscale - Phases 1 and 2
Description: The Positive and Negative Syndrome Scale (PANSS) will be used to measure symptom severity in this trial. PANSS is a 30-item questionnaire used to evaluate schizophrenia symptoms, based on the clinical interview as well as reports of family members or primary care hospital workers. PANSS consists of Positive scale (7 items), Negative scale (7 items), and General Psychopathological scale (16 items) sections. Each item (symptom) will be scored on a 7-point scale with higher scores representing increasing levels of psychopathology: 1) Absent, 2) Minimal, 3) Mild, 4) Moderate, 5) Moderate severe, 6) Severe, and 7) Extreme. Negative scale: 7 Items, (minimum score = 7, maximum score = 49)
Time Frame: Phase 1 timeframe is Day 0 and Day 14; Phase 2 timeframe is Day 14 and Day 28
Population: Ph 1 analysis includes the 34 subjects with Baseline PANSS data in the Placebo-Placebo (N=18) and Placebo-Drug (N=16) groups and 18 Drug-Drug group subjects. Per SPCD, the Ph 2 data excludes the 18 Drug-Drug group subjects and includes the 14 subjects in the Placebo-Drug group and 18 subjects in the Placebo-Placebo group with PANSS Baseline data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo - Placebo: Phase 1 - intravenous dextrose Phase 2 - intravenous dextrose
  Placebo:
Arm/Group | Drug | Placebo - Placebo
Number analyzed (Participants) | 32 | 34
units on a scale
  Phase 1 - Negative Score - Baseline: number analyzed (Participants) | 18 | 34
  Phase 1 - Negative Score - Baseline | 20.8 (5.8) | 20.6 (4.8)
  Phase 1 - Negative Score - Day 14: number analyzed (Participants) | 18 | 32
  Phase 1 - Negative Score - Day 14 | 19.0 (4.6) | 19.7 (5.1)
  Phase 1 - Negative Score - Change: number analyzed (Participants) | 18 | 32
  Phase 1 - Negative Score - Change | -1.8 (4.1) | -1.0 (2.8)
  Phase 2 - Negative Score - Day 14: number analyzed (Participants) | 14 | 18
  Phase 2 - Negative Score - Day 14 | 18.5 (5.8) | 20.7 (4.4)
  Phase 2 - Negative Score - Day 28: number analyzed (Participants) | 12 | 18
  Phase 2 - Negative Score - Day 28 | 18.0 (6.2) | 19.8 (4.7)
  Phase 2 - Negative Score - Change: number analyzed (Participants) | 12 | 18
  Phase 2 - Negative Score - Change | -0.1 (0.9) | -0.9 (2.9)
Statistical Analysis 1: Comparison: Drug vs Placebo - Placebo; Test type: Superiority; p = 0.85, ANCOVA; Mean Difference (Final Values) = -0.12
Statistical Analysis 2: Comparison: Drug vs Placebo - Placebo; Test type: Superiority; p = 0.88, ANCOVA; Mean Difference (Final Values) = -0.10

4. Secondary Outcome: PANSS - General Psychopathology Subscale - Phases 1 and 2
Description: The Positive and Negative Syndrome Scale (PANSS) will be used to measure symptom severity in this trial. PANSS is a 30-item questionnaire used to evaluate schizophrenia symptoms, based on the clinical interview as well as reports of family members or primary care hospital workers. PANSS consists of Positive scale (7 items), Negative scale (7 items), and General Psychopathological scale (16 items) sections. Each item (symptom) will be scored on a 7-point scale with higher scores representing increasing levels of psychopathology: 1) Absent, 2) Minimal, 3) Mild, 4) Moderate, 5) Moderate severe, 6) Severe, and 7) Extreme. General Psychopathology Subscale: 16 Items, (minimum score = 16, maximum score = 112)
Time Frame: Phase 1 timeframe is Baseline and Day 14; Phase 2 timeframe is Day 14 and Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug | Placebo - Placebo
Number analyzed (Participants) | 32 | 34
units on a scale
  Phase 1 - General Score - Baseline: number analyzed (Participants) | 18 | 34
  Phase 1 - General Score - Baseline | 37.6 (6.0) | 36.4 (5.1)
  Phase 1 - General Score - Day 14: number analyzed (Participants) | 18 | 32
  Phase 1 - General Score - Day 14 | 35.3 (7.1) | 35.5 (6.4)
  Phase 1 - General Score - Change: number analyzed (Participants) | 18 | 32
  Phase 1 - General Score - Change | -2.2 (7.0) | -0.6 (3.9)
  Phase 2 - General Score - Day 14: number analyzed (Participants) | 14 | 18
  Phase 2 - General Score - Day 14 | 34.7 (6.4) | 36.2 (6.6)
  Phase 2 - General Score - Day 28: number analyzed (Participants) | 12 | 18
  Phase 2 - General Score - Day 28 | 32.4 (5.6) | 32.4 (5.3)
  Phase 2 - General Score - Change: number analyzed (Participants) | 12 | 18
  Phase 2 - General Score - Change | -2.1 (5.2) | -3.7 (4.5)
Statistical Analysis 1: Comparison: Drug vs Placebo - Placebo; Test type: Superiority; p = 0.86, ANCOVA; Mean Difference (Final Values) = -0.19
Statistical Analysis 2: Comparison: Drug vs Placebo - Placebo; Test type: Superiority; p = 0.83, ANCOVA; Mean Difference (Final Values) = -0.23

5. Secondary Outcome: Average Percent Change From Baseline in the PANSS Total Score After 2 Weeks of Treatment Using SPCD
Description: as for outcome 1
Time Frame: For Phase 1, timeframe is Baseline and Day 14; Phase 2 timeframe is Day 14 and Day 28
Population: Ph 1 analysis includes 34 subjects with Baseline PANSS data in the Placebo-Placebo (N=18) and Placebo-Drug (N=16) groups and 18 Drug-Drug group subjects. Per SPCD, the Ph 2 data excludes 18 subjects in the Drug-Drug group and includes the 14 subjects in the Placebo-Drug group and 18 subjects in the Placebo-Placebo group with PANSS Baseline data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 32 | 34
percent change
  Phase 1 Average Percent Change from Baseline: number analyzed (Participants) | 18 | 34
  Phase 1 Average Percent Change from Baseline | -6.7 (12.8) | -3.2 (9.0)
  Phase 2 Average Percentage Change from Day 14: number analyzed (Participants) | 14 | 18
  Phase 2 Average Percentage Change from Day 14 | -3.0 (10.5) | -3.3 (8.1)

6. Secondary Outcome: Percentage of Subjects With 20% or More Reduction From Baseline in PANSS Total Score After 2 Weeks of Treatment Using SPCD
Description: as for outcome 1
Time Frame: For Phase 1, timeframe is Baseline and Day 14; Phase 2 timeframe is Day 14 and Day 28
Population: Phase 1 analysis combines the 34 subjects assigned to Placebo-Placebo (N=18) and Placebo-Drug (N=16) groups and the 18 subjects assigned to the Drug-Drug group with complete data at all visits. Per SPCD, the Phase 2 data includes the 14 subjects in the Placebo-Drug group and 18 subjects in the Placebo-Placebo group with complete data at all visits.
Measure: Number; unit: percent of subjects
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 32 | 34
percent of subjects
  Phase 1 % of subjects with >=20% reduction: number analyzed (Participants) | 18 | 34
  Phase 1 % of subjects with >=20% reduction | 16.67 | 0
  Phase 2 % of subjects with >=20% reduction: number analyzed (Participants) | 14 | 18
  Phase 2 % of subjects with >=20% reduction | 0 | 5.56

7. Secondary Outcome: Average Percent Change From Baseline in the PANSS Positive Subscale Score After 2 Weeks of Treatment Using SPCD
Description: The Positive and Negative Syndrome Scale (PANSS) will be used to measure symptom severity in this trial. PANSS is a 30-item questionnaire used to evaluate schizophrenia symptoms, based on the clinical interview as well as reports of family members or primary care hospital workers. PANSS consists of Positive scale (7 items), Negative scale (7 items), and General Psychopathological scale (16 items) sections. Each item (symptom) will be scored on a 7-point scale with higher scores representing increasing levels of psychopathology: 1) Absent, 2) Minimal, 3) Mild, 4) Moderate, 5) Moderate severe, 6) Severe, and 7) Extreme. Positive subscore scale: 7 items (minimum score = 7; maximum score = 49)
Time Frame: For Phase 1, timeframe is Baseline and Day 14; Phase 2 timeframe is Day 14 and Day 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 32 | 34
percent change
  Phase 1 Average Percent Change from Baseline: number analyzed (Participants) | 18 | 34
  Phase 1 Average Percent Change from Baseline | -7.9 (8.1) | -3.2 (13.6)
  Phase 2 Average Percentage Change from Day 14: number analyzed (Participants) | 14 | 18
  Phase 2 Average Percentage Change from Day 14 | -3.5 (15.4) | -2.9 (12.5)

8. Secondary Outcome: Average Percent Change From Baseline in the PANSS Negative Subscale Score After 2 Weeks of Treatment Using SPCD
Description: The Positive and Negative Syndrome Scale (PANSS) will be used to measure symptom severity in this trial. PANSS is a 30-item questionnaire used to evaluate schizophrenia symptoms, based on the clinical interview as well as reports of family members or primary care hospital workers. PANSS consists of Positive scale (7 items), Negative scale (7 items), and General Psychopathological scale (16 items) sections. Each item (symptom) will be scored on a 7-point scale with higher scores representing increasing levels of psychopathology: 1) Absent, 2) Minimal, 3) Mild, 4) Moderate, 5) Moderate severe, 6) Severe, and 7) Extreme. Negative subscore scale: 7 items (minimum score = 7; maximum score = 49)
Time Frame: For Phase 1, timeframe is Baseline and Day 14; Phase 2 timeframe is Day 14 and Day 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 32 | 34
percent change
  Phase 1 Average Percent Change from Baseline: number analyzed (Participants) | 18 | 34
  Phase 1 Average Percent Change from Baseline | -7.1 (17.6) | -4.6 (14.9)
  Phase 2 Average Percentage Change from Day 14: number analyzed (Participants) | 14 | 18
  Phase 2 Average Percentage Change from Day 14 | -7.9 (12.3) | -2.1 (16.5)

9. Secondary Outcome: Average Percent Change From Baseline in the PANSS General Psychopathology Subscale Score After 2 Weeks of Treatment Using SPCD
Description: The Positive and Negative Syndrome Scale (PANSS) will be used to measure symptom severity in this trial. PANSS is a 30-item questionnaire used to evaluate schizophrenia symptoms, based on the clinical interview as well as reports of family members or primary care hospital workers. PANSS consists of Positive scale (7 items), Negative scale (7 items), and General Psychopathological scale (16 items) sections. Each item (symptom) will be scored on a 7-point scale with higher scores representing increasing levels of psychopathology: 1) Absent, 2) Minimal, 3) Mild, 4) Moderate, 5) Moderate severe, 6) Severe, and 7) Extreme. General Psychopathology subscore scale: 16 items (minimum score = 16; maximum score = 112)
Time Frame: For Phase 1, timeframe is Baseline and Day 14; Phase 2 timeframe is Day 14 and Day 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 32 | 34
percent change
  Phase 1 Average Percent Change from Baseline: number analyzed (Participants) | 18 | 34
  Phase 1 Average Percent Change from Baseline | -4.8 (18.3) | -1.8 (10.9)
  Phase 2 Average Percentage Change from Day 14: number analyzed (Participants) | 14 | 18
  Phase 2 Average Percentage Change from Day 14 | 0.47 (13.3) | -3.7 (8.7)

10. Other Pre Specified Outcome: Change in the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) - Phases 1 and 2
Description: MATRICS: The Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB). The MATRICS Consensus Cognitive Battery is the standard tool for assessing cognitive change in trials of cognitive-enhancing agents in schizophrenia. The MCCB domains include: Speed of Processing; Attention/Vigilance; Working Memory; Verbal Learning; Visual Learning; Reasoning & Problem-Solving; and Social Cognition and the battery takes about 80 minutes to complete. The MCCB composite score represents a global measure of cognition. MCCB composite T scores are between 40 and 60 (normal range) and < 40 (below normal range).
Time Frame: Phase 1 timeframe is Baseline and Day 14; Phase 2 timeframe is Day 14 and Day 28
Population: Ph1 analysis includes 34 subjects with Baseline MATRICS data in the Placebo-Placebo (N=18) and Placebo-Drug (N=16) groups and 18 subjects the Drug-Drug group. Per SPCD, Ph 2 excludes the 18 subjects in the Drug-Drug group and includes the 14 subjects in the Placebo-Drug group and 18 subjects in the Placebo-Placebo group with Baseline MATRICS data.
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Drug | Placebo - Placebo
Number analyzed (Participants) | 32 | 34
T-scores
  Phase 1 - Baseline: number analyzed (Participants) | 18 | 34
  Phase 1 - Baseline | 26.2 (14.3) | 26.5 (14.5)
  Phase 1 - Day 14: number analyzed (Participants) | 18 | 32
  Phase 1 - Day 14 | 29.3 (12.9) | 28.6 (16.2)
  Phase 1 - Change: number analyzed (Participants) | 18 | 32
  Phase 1 - Change | 3.1 (3.9) | 1.4 (5.1)
  Phase 2 - Day 14: number analyzed (Participants) | 14 | 18
  Phase 2 - Day 14 | 28.8 (12.8) | 28.4 (18.8)
  Phase 2 - Day 28: number analyzed (Participants) | 12 | 18
  Phase 2 - Day 28 | 30.3 (13.6) | 31.0 (18.0)
  Phase 2 - Change: number analyzed (Participants) | 12 | 18
  Phase 2 - Change | 3.3 (4.2) | 2.6 (5.2)
Statistical Analysis 1: Comparison: Drug vs Placebo - Placebo; Test type: Superiority; p = 0.33, ANCOVA; Mean Difference (Final Values) = 1.12
Statistical Analysis 2: Comparison: Drug vs Placebo - Placebo; Test type: Superiority; p = 0.34, ANCOVA; Mean Difference (Final Values) = 1.10

11. Other Pre Specified Outcome: Average AIMS Total Scores (Items 1-7) by Group and Timepoint
Description: Abnormal Involuntary Movement Scale (AIMS):
  The AIMS Total Dyskinesia Score was calculated by averaging the first 7 items of the AIMS. The 7 items included in the AIMS Dyskinesia Score are rated on a scale from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score ranges from 0 to 4; a higher score reflects increased severity.
Time Frame: Baseline 1 (Day -1), 7 Hours Post-Infusion 1, Baseline 2 (Day 13), 7 Hours Post-Infusion 2, Final Follow-Up, including early termination visits
Population: Includes all subjects with AIMS data at Phases 1 and 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 16 | 18
units on a scale
  Baseline 1 | 0.72 (1.41) | 0.56 (0.96) | 0.56 (0.96)
  7 Hours Post-Infusion 1 | 0.56 (1.10) | 0.31 (0.48) | 0.31 (0.48)
  Baseline 2 | 0.44 (0.92) | 1.00 (1.47) | 1.00 (1.47)
  7 Hours Post-Infusion 2 | 0.47 (0.87) | 0.54 (0.88) | 0.54 (0.88)
  Final follow-up | 1.00 (2.09) | 0.93 (1.67) | 0.93 (1.67)

12. Other Pre Specified Outcome: Percent of Participants Rated as ≥ "Mild" or as "Yes" on AIMS Items 8-12
Description: Abnormal Involuntary Movement Scale (AIMS):
  The AIMS is a 12-item anchored score that is clinician administered and scored. Items are scored on a 0 (none) to 4 (severe) basis; items 8-10 deal with global severity; items 11-12 are yes-no questions concerning problems with teeth and/or dentures.
Time Frame: Baseline (Day -1), Follow-Up = reported at any assessment thereafter, including 7 hours after Infusions #1 and #2, Baseline 2 (Day 13) and final follow-up, including early termination visits.
Population: For each item, percentages of participants rated as exhibiting behaviors at the "mild" level or higher, or for items 11 and 12, as being present versus not (yes/no rated) are provided per treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 16 | 18
percentage of participants
  Baseline - Overall Severity Index (Item 8) | 5.6 | 6.3 | 11.1
  Follow-Up - Overall Severity Index (Item 8) | 16.7 | 18.8 | 16.7
  Baseline - Incapacitation (Item 9) | 0.0 | 0.0 | 5.6
  Follow-Up - Incapacitation (Item 9) | 0.0 | 6.3 | 0.0
  Baseline - Awareness (Item 10) | 11.1 | 6.3 | 5.6
  Follow-Up - Awareness (Item 10) | 5.6 | 18.8 | 5.6
  Baseline - Dental Problem (Item 11; % yes) | 22.2 | 31.3 | 16.7
  Follow-Up - Dental Problem (Item 11; % yes) | 27.8 | 37.5 | 22.2
  Baseline - Dentures (Item 12; % yes) | 5.6 | 18.8 | 16.7
  Follow-Up - Dentures (Item 12; % yes) | 11.1 | 31.3 | 22.2

13. Other Pre Specified Outcome: Change in The University of California San Diego (UCSD) Performance-based Skills Assessment Brief (UPSA-B) - Phases 1 and 2
Description: The University of California San Diego (UCSD) Performance-based Skills Assessment Brief (UPSA-B) consists of two of the five original UPSA domains, finances and communication. Each subscale contributes 50 points; total scores range from 0 to 100 points with higher scores reflecting better performance.
Time Frame: Phase 1 timeframe is Baseline and Day 14; Phase 2 timeframe is Day 14 and Day 28
Population: Ph1 analysis includes 34 subjects with Baseline UPSA-B data in the Placebo-Placebo (N=18) and Placebo-Drug (N=16) groups and 18 subjects the Drug-Drug group. Per SPCD, Ph 2 excludes the 18 subjects in the Drug-Drug group and includes the 14 subjects in the Placebo-Drug group and 18 subjects in the Placebo-Placebo group with Baseline UPSA-B data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug | Placebo - Placebo
Number analyzed (Participants) | 32 | 34
units on a scale
  Phase 1 - Baseline: number analyzed (Participants) | 18 | 34
  Phase 1 - Baseline | 74.0 (17.2) | 71.8 (17.1)
  Phase 1 - Day 14: number analyzed (Participants) | 18 | 32
  Phase 1 - Day 14 | 76.7 (17.4) | 77.9 (14.6)
  Phase 1 - Change: number analyzed (Participants) | 18 | 32
  Phase 1 - Change | 2.7 (7.6) | 6.2 (9.9)
  Phase 2 - Day 14: number analyzed (Participants) | 14 | 18
  Phase 2 - Day 14 | 80.2 (13.1) | 76.0 (15.9)
  Phase 2 - Day 28: number analyzed (Participants) | 12 | 18
  Phase 2 - Day 28 | 85.4 (11.2) | 74.5 (20.9)
  Phase 2 - Change: number analyzed (Participants) | 12 | 18
  Phase 2 - Change | 5.5 (7.7) | -1.5 (10.9)
Statistical Analysis 1: Comparison: Drug vs Placebo - Placebo; Test type: Superiority; p = 0.34, ANCOVA; Mean Difference (Final Values) = 1.11
Statistical Analysis 2: Comparison: Drug vs Placebo - Placebo; Test type: Superiority; p = 0.36, ANCOVA; Mean Difference (Final Values) = 2.05

14. Other Pre Specified Outcome: Number of Participants Reporting Suicidal Ideation/Behavior on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia Suicide Severity Rating Scale (C-SSRS): The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed in the National Institute of Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment. It is a clinical interview providing a summary of both ideation and behavior that can be administered during any evaluation or risk assessment to identify the level and type of suicidality present. The C-SSRS can also be used during treatment to monitor for clinical worsening or improvement. It contains 5 rating scale questions (yes/no) for suicidal ideation increasing severity and 5 rating scale questions (yes/no) for suicidal behavior of increasing severity. The time frame is for both lifetime and the past six months for the Baseline/Screening scale and since the last visit for the Since Last Visit scale.
Time Frame: Screening Visit, Days 3 (Baseline 1), Days 7, 13 (Baseline 2), 21 and 28
Population: All subjects with C-SSRS data reporting suicidal ideation/behavior
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
Number analyzed (Participants) | 23 | 19 | 18
Participants
  Suicidal ideation (SI) (% any of the following) | 2 | 1 | 2
  Wish to be dead | 1 | 1 | 1
  Non-specific active suicidal thoughts | 2 | 1 | 1
  Active SI w/any method (no plan) W/O intent to act | 0 | 0 | 0
  Active SI w/some intent to act, W/O specific plan | 0 | 0 | 0
  Active SI with specific plan & intent | 0 | 0 | 0
  Suicidal behavior (% any of the following) | 0 | 0 | 0
  Prepatory acts or behavior | 0 | 0 | 0
  Aborted attempt | 0 | 0 | 0
  Interrupted attempt | 0 | 0 | 0
  Non-fatal suicide attempt | 0 | 0 | 0
  Self-injurious behavior W/O suicidal intent | 0 | 0 | 0

15. Other Pre Specified Outcome: Systolic Blood Pressure Per Infusion Phase by Group
Description: Infusion 1 (Day 0) - Systolic Blood Pressure at all time points by group
  "Phase" in this analysis refers to the infusion stage as defined in the protocol.
Time Frame: Day 0 - Phase 1 - Baseline = min000s1 and @5 min; Phase 2 - Baseline = min000 then every 10 minutes for 4 hours; Post Infusion - Baseline = min000, then every 10 minutes for 2 hours
Population: Includes all subjects during Phase 1 (i.e., infusion 1)
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Drug-Drug: Phase 1 - intravenous sodium nitroprusside Phase 2 - intravenous sodium nitroprusside
  sodium nitroprusside: intravenous
- Placebo-Drug: Phase 1 - intravenous dextrose Phase 2 - intravenous sodium nitroprusside
Arm/Group | Drug-Drug | Placebo-Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 16 | 18
mmHg
  Phase 1 - min000s1 | 121.79 (14.46) | 121.50 (10.65) | 123.78 (11.46)
  Phase 1 - min005s1 | 116.95 (12.78) | 126.13 (13.01) | 121.94 (14.39)
  Phase 2 - min000 | 114.89 (13.13) | 125.13 (11.04) | 121.00 (12.86)
  Phase 2 - min005: number analyzed (Participants) | 14 | 16 | 18
  Phase 2 - min005 | 111.32 (11.51) | 124.38 (10.29) | 121.00 (14.12)
  Phase 2 - min010: number analyzed (Participants) | 14 | 16 | 18
  Phase 2 - min010 | 112.72 (12.84) | 127.06 (8.93) | 122.33 (11.56)
  Phase 2 - min015: number analyzed (Participants) | 14 | 16 | 18
  Phase 2 - min015 | 111.28 (9.48) | 125.75 (10.51) | 121.94 (11.58)
  Phase 2 - min020 | 108.28 (10.21) | 124.63 (9.94) | 121.11 (10.81)
  Phase 2 - min025 | 109.83 (10.70) | 126.63 (11.89) | 121.11 (11.80)
  Phase 2 - min030 | 108.61 (10.01) | 125.13 (9.84) | 119.67 (13.77)
  Phase 2 - min040 | 111.82 (9.80) | 125.63 (11.86) | 122.56 (11.46)
  Phase 2 - min050 | 111.00 (8.89) | 125.73 (9.32) | 122.56 (11.46)
  Phase 2 - min060 | 112.53 (11.99) | 126.87 (9.69) | 120.17 (12.91)
  Phase 2 - min070 | 114.82 (12.83) | 126.27 (8.86) | 120.11 (10.76)
  Phase 2 - min080 | 110.00 (9.98) | 125.53 (9.62) | 120.83 (13.90)
  Phase 2 - min090 | 111.94 (9.83) | 125.00 (11.14) | 121.33 (12.88)
  Phase 2 - min100 | 111.00 (12.97) | 123.87 (11.75) | 122.11 (12.39)
  Phase 2 - min110 | 112.29 (7.83) | 128.33 (10.60) | 122.83 (12.32)
  Phase 2 - min120 | 111.76 (10.56) | 124.93 (12.57) | 119.06 (15.30)
  Phase 2 - min130 | 109.82 (9.19) | 125.20 (8.99) | 119.17 (10.63)
  Phase 2 - min140 | 109.47 (7.34) | 127.67 (9.76) | 119.72 (11.20)
  Phase 2 - min150 | 110.12 (9.62) | 126.93 (10.75) | 123.39 (12.95)
  Phase 2 - min160 | 107.88 (9.97) | 126.00 (9.56) | 121.72 (15.23)
  Phase 2 - min170 | 109.35 (11.89) | 124.33 (9.51) | 122.72 (15.14)
  Phase 2 - min180 | 110.06 (9.85) | 127.07 (12.63) | 123.22 (13.01)
  Phase 2 - min190 | 110.12 (11.60) | 125.13 (13.10) | 121.94 (12.46)
  Phase 2 - min200 | 107.41 (12.57) | 125.40 (13.00) | 122.67 (14.63)
  Phase 2 - min210 | 109.71 (8.08) | 131.87 (13.79) | 122.94 (11.34)
  Phase 2 - min220 | 109.82 (9.57) | 125.73 (13.24) | 125.89 (14.58)
  Phase 2 - min230 | 109.35 (9.57) | 126.00 (13.80) | 124.61 (13.75)
  Phase 2 - min240 | 109.53 (9.13) | 128.67 (14.01) | 124.44 (14.16)
  Post Infusion - min000 | 107.50 (11.53) | 128.38 (13.87) | 125.22 (13.80)
  Post Infusion - min005 | 114.44 (11.01) | 126.13 (13.84) | 123.12 (10.01)
  Post Infusion - min010 | 116.28 (11.74) | 127.33 (12.80) | 122.06 (11.62)
  Post Infusion - min015 | 117.22 (11.07) | 128.40 (16.79) | 124.67 (11.96)
  Post Infusion - min020 | 117.39 (9.12) | 128.80 (13.04) | 124.50 (12.08)
  Post Infusion - min025 | 116.33 (12.58) | 129.53 (14.94) | 126.72 (14.74)
  Post Infusion - min030 | 118.56 (11.93) | 129.81 (13.96) | 124.00 (14.12)
  Post Infusion - min040 | 119.67 (12.03) | 128.33 (14.99) | 123.33 (14.48)
  Post Infusion - min050 | 117.33 (13.91) | 128.47 (11.86) | 123.11 (13.78)
  Post Infusion - min060 | 122.22 (12.35) | 129.93 (12.21) | 124.61 (14.97)
  Post Infusion - min070 | 122.33 (13.78) | 130.27 (11.51) | 122.72 (15.86)
  Post Infusion - min080 | 118.83 (12.78) | 128.47 (11.86) | 122.94 (14.49)
  Post Infusion - min090 | 117.67 (12.56) | 129.20 (13.03) | 124.06 (10.94)
  Post Infusion - min100 | 120.44 (11.87) | 125.67 (11.63) | 121.72 (10.65)
  Post Infusion - min110 | 122.61 (13.42) | 129.27 (11.49) | 125.06 (14.58)
  Post Infusion - min120 | 122.22 (13.41) | 128.67 (10.99) | 124.44 (12.34)

16. Other Pre Specified Outcome: Diastolic Blood Pressure Per Infusion Phase by Group
Description: Infusion 1 (Day 0) - Diastolic Blood Pressure at all time points by group
  "Phase" in this analysis refers to the infusion stage as defined in the protocol.
Time Frame: as for outcome 15
Population: Includes all subjects during Phase 1 (i.e., infusion 1)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Drug-Drug | Placebo-Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 16 | 18
mmHg
  Phase 1 - min000s1 | 71.63 (19.03) | 75.13 (10.44) | 75.11 (10.12)
  Phase 1 - min005s1 | 68.79 (10.12) | 75.38 (6.30) | 74.94 (9.91)
  Phase 2 - min000 | 67.58 (10.18) | 74.44 (7.28) | 74.72 (11.88)
  Phase 2 - min005 | 66.37 (12.88) | 74.31 (7.01) | 74.39 (8.42)
  Phase 2 - min010 | 65.72 (14.70) | 75.50 (8.09) | 73.72 (9.50)
  Phase 2 - min015 | 62.67 (9.94) | 74.75 (8.38) | 72.78 (8.61)
  Phase 2 - min020 | 62.06 (9.33) | 75.19 (8.29) | 74.33 (12.25)
  Phase 2 - min025 | 62.33 (8.61) | 74.31 (6.02) | 72.83 (11.20)
  Phase 2 - min030 | 60.78 (8.93) | 75.50 (8.09) | 72.06 (11.67)
  Phase 2 - min040 | 61.29 (7.46) | 75.06 (9.76) | 72.67 (11.66)
  Phase 2 - min050 | 60.65 (7.52) | 76.47 (10.23) | 71.28 (10.06)
  Phase 2 - min060 | 61.88 (9.50) | 75.80 (9.30) | 71.94 (11.11)
  Phase 2 - min070 | 64.53 (11.21) | 75.27 (9.62) | 71.11 (12.74)
  Phase 2 - min080 | 62.41 (10.89) | 76.73 (9.80) | 71.61 (11.69)
  Phase 2 - min090 | 64.18 (11.48) | 74.53 (9.81) | 73.11 (14.06)
  Phase 2 - min100 | 62.29 (8.96) | 74.87 (7.74) | 73.94 (11.50)
  Phase 2 - min110 | 63.94 (6.97) | 77.07 (12.02) | 72.06 (12.98)
  Phase 2 - min120 | 66.94 (12.02) | 74.20 (8.94) | 72.28 (14.71)
  Phase 2 - min130 | 62.47 (8.87) | 76.27 (8.44) | 69.72 (13.47)
  Phase 2 - min140 | 61.94 (8.75) | 78.27 (8.96) | 71.06 (10.98)
  Phase 2 - min150 | 64.53 (6.38) | 75.60 (8.10) | 73.83 (11.74)
  Phase 2 - min160 | 61.88 (8.99) | 75.53 (17.01) | 72.22 (10.50)
  Phase 2 - min170 | 62.29 (6.28) | 74.40 (9.30) | 72.83 (11.74)
  Phase 2 - min180 | 62.06 (9.05) | 74.20 (9.67) | 72.22 (12.74)
  Phase 2 - min190 | 63.47 (9.41) | 74.67 (7.48) | 73.56 (11.93)
  Phase 2 - min200 | 64.18 (7.57) | 78.60 (9.83) | 74.33 (11.63)
  Phase 2 - min210 | 63.82 (9.51) | 76.20 (8.83) | 75.56 (11.22)
  Phase 2 - min220 | 63.47 (10.40) | 76.00 (9.06) | 75.17 (12.94)
  Phase 2 - min230 | 60.82 (9.13) | 76.40 (7.95) | 74.17 (9.82)
  Phase 2 - min240 | 63.47 (8.46) | 76.53 (7.79) | 74.00 (10.19)
  Post Infusion - min000 | 62.56 (8.69) | 77.50 (8.40) | 74.67 (11.11)
  Post Infusion - min005 | 67.17 (9.67) | 76.40 (8.49) | 76.18 (9.19)
  Post Infusion - min010 | 66.78 (9.90) | 78.07 (9.03) | 75.56 (13.17)
  Post Infusion - min015 | 69.00 (10.84) | 76.20 (9.65) | 75.78 (11.33)
  Post Infusion - min020 | 71.72 (11.10) | 77.80 (12.25) | 75.61 (12.53)
  Post Infusion - min025 | 66.72 (11.40) | 78.87 (10.80) | 77.06 (10.80)
  Post Infusion - min030 | 69.67 (9.00) | 78.81 (9.70) | 75.33 (11.75)
  Post Infusion - min040 | 68.06 (11.43) | 77.53 (10.85) | 75.89 (11.84)
  Post Infusion - min050 | 69.56 (10.78) | 78.40 (7.27) | 75.17 (11.81)
  Post Infusion - min060 | 68.83 (10.44) | 79.33 (11.17) | 74.61 (10.87)
  Post Infusion - min070 | 70.22 (10.33) | 78.13 (7.49) | 75.28 (9.37)
  Post Infusion - min080 | 71.89 (10.02) | 76.60 (7.49) | 75.06 (13.17)
  Post Infusion - min090 | 69.89 (7.08) | 79.07 (9.06) | 74.44 (10.07)
  Post Infusion - min100 | 69.50 (9.24) | 76.80 (10.75) | 73.56 (10.61)
  Post Infusion - min110 | 71.61 (8.13) | 76.53 (10.64) | 74.22 (9.74)
  Post Infusion - min120 | 70.61 (9.86) | 78.27 (8.40) | 75.89 (8.53)

17. Other Pre Specified Outcome: Systolic Blood Pressure Per Infusion Phase by Group
Description: Infusion 2 (Day 14) - Systolic Blood Pressure at all time points by group
  "Phase" in this analysis refers to the infusion stage as defined in the protocol.
Time Frame: Day 14 - Phase 1 - Baseline = min000s1 and @5 min; Phase 2 - Baseline = min000 then every 10 minutes for 4 hours; Post Infusion - Baseline = min000, then every 10 minutes for 2 hours
Population: Includes all subjects during Phase 2 (i.e., infusion 2)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Drug-Drug | Placebo-Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 14 | 18
mmHg
  Phase 1 - min000s1 | 120.69 (11.84) | 121.92 (9.66) | 122.61 (10.22)
  Phase 1 - min005s1 | 112.69 (12.38) | 120.77 (12.38) | 119.39 (10.67)
  Phase 2 - min000 | 110.88 (11.61) | 120.92 (14.20) | 120.78 (12.08)
  Phase 2 - min005 | 107.50 (11.36) | 116.31 (9.96) | 120.39 (12.22)
  Phase 2 - min010 | 108.50 (9.39) | 113.38 (12.53) | 120.41 (12.62)
  Phase 2 - min015 | 108.88 (9.06) | 113.46 (10.32) | 117.28 (13.35)
  Phase 2 - min020 | 108.19 (8.93) | 112.62 (10.66) | 117.94 (12.65)
  Phase 2 - min025 | 110.81 (11.11) | 115.62 (13.88) | 118.22 (14.40)
  Phase 2 - min030 | 109.88 (8.43) | 113.69 (16.09) | 116.44 (13.40)
  Phase 2 - min040 | 108.06 (8.46) | 117.54 (16.58) | 118.94 (11.57)
  Phase 2 - min050 | 109.00 (10.22) | 112.77 (13.91) | 118.56 (15.60)
  Phase 2 - min060 | 109.63 (13.20) | 113.31 (14.12) | 116.94 (12.75)
  Phase 2 - min070 | 108.56 (10.46) | 113.15 (12.15) | 118.50 (14.20)
  Phase 2 - min080 | 108.50 (10.98) | 113.08 (15.34) | 118.50 (13.57)
  Phase 2 - min090 | 109.06 (10.59) | 109.00 (11.63) | 118.06 (12.49)
  Phase 2 - min100 | 106.94 (11.58) | 111.50 (16.10) | 119.00 (14.98)
  Phase 2 - min110 | 105.67 (7.80) | 112.46 (16.04) | 120.39 (11.95)
  Phase 2 - min120 | 105.87 (9.19) | 106.33 (10.87) | 118.83 (15.25)
  Phase 2 - min130 | 108.53 (10.70) | 110.17 (11.75) | 120.06 (13.58)
  Phase 2 - min140 | 111.27 (10.50) | 110.54 (11.23) | 120.33 (15.11)
  Phase 2 - min150 | 112.13 (11.42) | 110.83 (18.52) | 117.67 (12.76)
  Phase 2 - min160 | 109.87 (11.11) | 116.17 (13.07) | 121.17 (13.79)
  Phase 2 - min170 | 114.33 (12.61) | 113.33 (12.04) | 120.61 (12.65)
  Phase 2 - min180 | 111.27 (9.38) | 113.92 (11.77) | 117.67 (11.44)
  Phase 2 - min190 | 110.47 (9.82) | 114.83 (16.46) | 120.72 (11.74)
  Phase 2 - min200 | 110.40 (13.47) | 115.08 (16.76) | 120.94 (14.24)
  Phase 2 - min210 | 113.13 (14.71) | 114.33 (17.85) | 121.17 (11.75)
  Phase 2 - min220 | 109.20 (15.18) | 112.33 (11.54) | 120.06 (11.44)
  Phase 2 - min230 | 110.27 (12.79) | 113.58 (12.92) | 118.83 (12.64)
  Phase 2 - min240 | 108.53 (9.48) | 111.83 (12.58) | 119.00 (12.29)
  Post Infusion - min000 | 107.75 (9.94) | 113.25 (13.51) | 118.22 (120.28)
  Post Infusion - min005 | 111.06 (12.41) | 118.25 (18.23) | 120.28 (11.93)
  Post Infusion - min010 | 116.88 (16.70) | 122.83 (16.03) | 122.94 (10.91)
  Post Infusion - min015 | 114.75 (15.07) | 124.58 (16.14) | 122.78 (11.70)
  Post Infusion - min020 | 115.00 (11.55) | 122.92 (13.24) | 121.56 (12.60)
  Post Infusion - min025 | 116.00 (12.41) | 125.83 (16.94) | 126.67 (15.06)
  Post Infusion - min030 | 117.50 (12.56) | 123.67 (16.54) | 126.06 (14.86)
  Post Infusion - min040 | 118.44 (11.40) | 123.92 (11.24) | 122.11 (13.75)
  Post Infusion - min050 | 122.75 (22.66) | 124.17 (13.19) | 122.72 (14.82)
  Post Infusion - min060 | 125.31 (14.93) | 121.08 (12.45) | 123.17 (15.00)
  Post Infusion - min070 | 122.44 (19.68) | 120.33 (10.46) | 124.78 (14.82)
  Post Infusion - min080 | 122.38 (15.21) | 121.83 (14.65) | 123.17 (13.34)
  Post Infusion - min090 | 122.25 (14.19) | 125.08 (13.73) | 126.28 (14.52)
  Post Infusion - min100 | 121.94 (21.68) | 123.92 (10.99) | 122.94 (16.25)
  Post Infusion - min110 | 123.50 (13.57) | 125.17 (16.51) | 125.06 (11.88)
  Post Infusion - min120 | 122.31 (16.41) | 125.75 (12.26) | 125.00 (12.29)

18. Other Pre Specified Outcome: Phase 2 - Diastolic Blood Pressure Per Infusion Phase by Group
Description: Infusion 2 (Day 14) - Diastolic Blood Pressure at all time points by group
Time Frame: as for outcome 17
Population: Includes all subjects during Phase 1 (i.e., infusion 1)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Drug-Drug | Placebo-Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 14 | 18
mmHg
  Phase 1 - min000s1 | 69.38 (7.80) | 74.50 (8.89) | 74.50 (8.89)
  Phase 1 - min005s1 | 63.56 (8.78) | 73.89 (8.70) | 73.89 (8.70)
  Phase 2 - min000 | 63.94 (8.46) | 72.72 (8.84) | 72.72 (8.84)
  Phase 2 - min005 | 61.00 (6.23) | 71.28 (7.28) | 71.28 (7.28)
  Phase 2 - min010 | 61.63 (7.57) | 74.65 (9.03) | 74.65 (9.03)
  Phase 2 - min015 | 61.44 (9.06) | 73.50 (7.15) | 73.50 (7.15)
  Phase 2 - min020 | 63.19 (8.72) | 70.94 (7.07) | 70.94 (7.07)
  Phase 2 - min025 | 59.25 (8.29) | 71.56 (9.10) | 71.56 (9.10)
  Phase 2 - min030 | 61.75 (7.87) | 71.11 (7.23) | 71.11 (7.23)
  Phase 2 - min040 | 59.94 (8.82) | 73.17 (9.07) | 73.17 (9.07)
  Phase 2 - min050 | 60.25 (8.42) | 71.89 (12.07) | 71.89 (12.07)
  Phase 2 - min060 | 60.38 (11.97) | 71.44 (12.23) | 71.44 (12.23)
  Phase 2 - min070 | 59.19 (10.78) | 71.00 (10.77) | 71.00 (10.77)
  Phase 2 - min080 | 59.00 (7.38) | 70.72 (12.81) | 70.72 (12.81)
  Phase 2 - min090 | 57.13 (7.83) | 70.22 (12.34) | 70.22 (12.34)
  Phase 2 - min100 | 58.13 (8.37) | 71.00 (12.39) | 71.00 (12.39)
  Phase 2 - min110 | 59.73 (5.97) | 71.89 (11.54) | 71.89 (11.54)
  Phase 2 - min120 | 59.47 (8.59) | 68.28 (10.65) | 68.28 (10.65)
  Phase 2 - min130 | 60.33 (8.16) | 73.44 (11.94) | 73.44 (11.94)
  Phase 2 - min140 | 58.73 (10.23) | 71.56 (10.87) | 71.56 (10.87)
  Phase 2 - min150 | 61.87 (10.10) | 74.06 (12.80) | 74.06 (12.80)
  Phase 2 - min160 | 60.53 (7.68) | 73.94 (10.41) | 73.94 (10.41)
  Phase 2 - min170 | 61.87 (11.60) | 74.61 (8.43) | 74.61 (8.43)
  Phase 2 - min180 | 60.27 (9.00) | 72.28 (8.17) | 72.28 (8.17)
  Phase 2 - min190 | 59.73 (10.23) | 73.00 (10.99) | 73.00 (10.99)
  Phase 2 - min200 | 58.40 (7.03) | 73.56 (10.35) | 73.56 (10.35)
  Phase 2 - min210 | 60.27 (9.00) | 74.11 (11.53) | 74.11 (11.53)
  Phase 2 - min220 | 59.13 (8.60) | 72.22 (9.62) | 72.22 (9.62)
  Phase 2 - min230 | 62.00 (8.12) | 72.33 (10.48) | 72.33 (10.48)
  Phase 2 - min240 | 59.60 (8.58) | 70.11 (8.05) | 70.11 (8.05)
  Post Infusion - min000 | 59.81 (8.42) | 70.39 (8.10) | 70.39 (8.10)
  Post Infusion - min005 | 63.31 (7.87) | 71.94 (9.14) | 71.94 (9.14)
  Post Infusion - min010 | 67.06 (9.26) | 73.39 (9.76) | 73.39 (9.76)
  Post Infusion - min015 | 65.13 (10.20) | 75.67 (10.79) | 75.67 (10.79)
  Post Infusion - min020 | 69.44 (12.44) | 74.89 (9.62) | 74.89 (8.66)
  Post Infusion - min025 | 66.88 (12.94) | 76.89 (8.66) | 76.89 (8.66)
  Post Infusion - min030 | 68.81 (12.45) | 76.89 (14.57) | 76.89 (14.57)
  Post Infusion - min040 | 70.31 (14.89) | 72.39 (11.32) | 72.39 (11.32)
  Post Infusion - min050 | 70.25 (10.79) | 74.72 (12.56) | 74.72 (12.56)
  Post Infusion - min060 | 67.69 (7.88) | 74.11 (11.90) | 74.11 (11.90)
  Post Infusion - min070 | 68.81 (9.72) | 76.78 (10.28) | 76.78 (10.28)
  Post Infusion - min080 | 68.88 (7.87) | 74.61 (11.25) | 74.61 (11.25)
  Post Infusion - min090 | 69.88 (8.87) | 73.83 (11.40) | 73.83 (11.40)
  Post Infusion - min100 | 69.38 (8.61) | 74.28 (12.15) | 74.28 (12.15)
  Post Infusion - min110 | 70.81 (9.09) | 77.11 (10.78) | 77.11 (10.78)
  Post Infusion - min120 | 70.56 (7.69) | 78.00 (9.15) | 78.00 (9.15)

19. Other Pre Specified Outcome: Heart Rate Per Infusion Phase by Group
Description: Infusion 1 (Day 0) - Heart rate at all time points by group
  "Phase" in this analysis refers to the infusion stage as defined in the protocol.
Time Frame: as for outcome 15
Population: Includes all subjects during Phase 1 (i.e., infusion 1)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Drug-Drug | Placebo-Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 16 | 18
bpm
  Phase 1 - min000s1 | 78.47 (13.11) | 79.00 (15.84) | 79.94 (17.67)
  Phase 1 - min005s1 | 81.21 (15.79) | 77.81 (14.39) | 79.44 (16.33)
  Phase 2 - min000 | 84.00 (13.81) | 76.94 (15.05) | 79.94 (16.86)
  Phase 2 - min005 | 85.47 (13.49) | 77.88 (15.13) | 78.00 (17.19)
  Phase 2 - min010 | 85.17 (13.44) | 77.25 (14.75) | 79.61 (16.75)
  Phase 2 - min015 | 84.33 (13.97) | 78.00 (14.01) | 77.89 (17.33)
  Phase 2 - min020 | 83.00 (13.84) | 76.44 (14.77) | 79.28 (17.28)
  Phase 2 - min025 | 83.83 (14.61) | 77.13 (13.61) | 77.06 (17.12)
  Phase 2 - min030 | 83.94 (14.21) | 76.69 (14.38) | 78.83 (17.57)
  Phase 2 - min040 | 83.06 (13.98) | 77.88 (14.42) | 77.56 (18.10)
  Phase 2 - min050 | 83.65 (14.28) | 76.67 (13.28) | 79.50 (18.06)
  Phase 2 - min060 | 83.59 (13.86) | 78.13 (12.88) | 78.56 (17.12)
  Phase 2 - min070 | 82.53 (13.73) | 77.07 (12.66) | 77.11 (17.27)
  Phase 2 - min080 | 84.76 (13.37) | 76.47 (15.08) | 76.89 (17.83)
  Phase 2 - min090 | 83.82 (12.73) | 77.80 (14.36) | 76.22 (17.13)
  Phase 2 - min100 | 84.29 (12.46) | 78.53 (12.82) | 75.94 (16.31)
  Phase 2 - min110 | 85.18 (12.54) | 76.73 (11.66) | 75.44 (16.76)
  Phase 2 - min120 | 83.71 (11.97) | 78.47 (13.52) | 78.39 (20.37)
  Phase 2 - min130 | 83.59 (12.50) | 77.33 (12.66) | 75.94 (15.69)
  Phase 2 - min140 | 81.76 (11.99) | 77.60 (12.79) | 75.28 (16.35)
  Phase 2 - min150 | 82.06 (13.38) | 79.67 (11.79) | 76.06 (15.42)
  Phase 2 - min160 | 83.41 (11.49) | 78.73 (11.81) | 79.33 (16.11)
  Phase 2 - min170 | 83.88 (11.19) | 79.07 (13.57) | 76.44 (18.07)
  Phase 2 - min180 | 82.12 (10.34) | 77.53 (13.72) | 78.56 (16.76)
  Phase 2 - min190 | 83.24 (12.40) | 79.40 (15.08) | 76.89 (16.36)
  Phase 2 - min200 | 83.41 (11.37) | 79.27 (13.42) | 80.00 (15.98)
  Phase 2 - min210 | 81.24 (11.68) | 80.27 (14.39) | 77.50 (15.57)
  Phase 2 - min220 | 82.94 (12.29) | 79.93 (14.10) | 77.33 (16.83)
  Phase 2 - min230 | 84.47 (12.96) | 79.87 (15.06) | 78.78 (16.75)
  Phase 2 - min240 | 85.29 (12.01) | 79.40 (13.74) | 78.56 (16.85)
  Post Infusion - min000 | 86.28 (11.96) | 82.44 (14.81) | 78.11 (16.91)
  Post Infusion - min005 | 80.39 (12.46) | 80.80 (15.81) | 80.29 (16.13)
  Post Infusion - min010 | 80.78 (12.74) | 78.67 (1317) | 78.83 (14.77)
  Post Infusion - min015 | 80.67 (10.32) | 79.93 (13.34) | 79.39 (15.79)
  Post Infusion - min020 | 82.06 (10.78) | 82.13 (13.91) | 80.33 (16.94)
  Post Infusion - min025 | 79.78 (11.83) | 81.60 (13.83) | 78.22 (17.13)
  Post Infusion - min030 | 79.39 (13.56) | 82.13 (13.07) | 79.72 (16.44)
  Post Infusion - min040 | 79.72 (12.55) | 81.47 (13.41) | 78.72 (15.97)
  Post Infusion - min050 | 79.06 (12.32) | 78.47 (13.45) | 81.28 (15.18)
  Post Infusion - min060 | 79.17 (11.93) | 79.40 (12.40) | 78.83 (15.96)
  Post Infusion - min070 | 79.83 (10.74) | 81.87 (15.81) | 79.94 (14.49)
  Post Infusion - min080 | 78.44 (10.92) | 83.87 (11.54) | 80.33 (16.22)
  Post Infusion - min090 | 79.11 (12.36) | 82.33 (12.82) | 79.22 (17.16)
  Post Infusion - min100 | 79.17 (12.66) | 84.67 (12.58) | 80.00 (16.95)
  Post Infusion - min110 | 79.67 (11.74) | 82.80 (13.61) | 80.61 (16.55)
  Post Infusion - min120 | 79.56 (11.98) | 83.47 (13.44) | 80.00 (16.37)

20. Other Pre Specified Outcome: Heart Rate Per Infusion Phase by Group
Description: Infusion 2 (Day 14) - Heart rate at all time points by group
  "Phase" in this analysis refers to the infusion stage as defined in the protocol.
Time Frame: as for outcome 17
Population: Includes all subjects during Phase 1 (i.e., infusion 1)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Drug-Drug | Placebo-Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 14 | 18
bpm
  Phase 1 - min000s1 | 77.38 (11.77) | 75.08 (13.94) | 76.94 (18.50)
  Phase 1 - min005s1 | 79.69 (12.43) | 76.77 (14.86) | 78.67 (17.85)
  Phase 2 - min000 | 81.06 (11.25) | 77.77 (15.24) | 78.72 (17.75)
  Phase 2 - min005 | 82.31 (12.88) | 81.38 (15.32) | 76.39 (17.77)
  Phase 2 - min010 | 81.50 (13.46) | 80.62 (16.44) | 77.12 (17.19)
  Phase 2 - min015 | 81.38 (12.99) | 80.92 (15.40) | 76.06 (17.11)
  Phase 2 - min020 | 82.06 (12.13) | 79.69 (16.73) | 74.89 (16.97)
  Phase 2 - min025 | 82.31 (12.35) | 80.69 (18.08) | 76.22 (16.81)
  Phase 2 - min030 | 81.50 (10.22) | 81.15 (16.32) | 76.17 (15.73)
  Phase 2 - min040 | 79.88 (13.61) | 81.69 (15.50) | 76.72 (15.35)
  Phase 2 - min050 | 80.25 (12.23) | 78.85 (15.42) | 75.00 (16.30)
  Phase 2 - min060 | 79.69 (15.12) | 79.69 (14.63) | 75.50 (15.75)
  Phase 2 - min070 | 81.69 (13.85) | 81.31 (13.53) | 75.06 (16.28)
  Phase 2 - min080 | 79.44 (13.93) | 80.23 (14.11) | 75.39 (14.61)
  Phase 2 - min090 | 78.00 (14.58) | 79.58 (14.71) | 73.78 (15.56)
  Phase 2 - min100 | 79.94 (14.29) | 78.17 (14.66) | 76.11 (15.15)
  Phase 2 - min110 | 83.33 (11.58) | 80.15 (15.51) | 75.17 (15.52)
  Phase 2 - min120 | 82.47 (12.97) | 81.25 (16.16) | 74.56 (14.27)
  Phase 2 - min130 | 82.13 (13.03) | 78.75 (15.24) | 75.11 (13.60)
  Phase 2 - min140 | 81.73 (13.95) | 80.69 (14.92) | 75.89 (15.87)
  Phase 2 - min150 | 81.40 (12.57) | 78.75 (13.59) | 75.78 (14.53)
  Phase 2 - min160 | 81.53 (13.20) | 80.00 (11.26) | 75.33 (13.75)
  Phase 2 - min170 | 81.60 (14.46) | 78.75 (12.55) | 75.06 (14.43)
  Phase 2 - min180 | 80.00 (12.91) | 81.25 (12.81) | 74.78 (14.10)
  Phase 2 - min190 | 80.93 (12.91) | 80.58 (16.37) | 73.94 (14.18)
  Phase 2 - min200 | 81.60 (14.39) | 80.33 (14.27) | 75.00 (12.63)
  Phase 2 - min210 | 84.73 (11.93) | 80.75 (17.12) | 75.33 (15.04)
  Phase 2 - min220 | 84.07 (12.55) | 79.92 (13.92) | 74.61 (14.46)
  Phase 2 - min230 | 85.07 (11.78) | 78.00 (14.59) | 77.56 (14.61)
  Phase 2 - min240 | 82.53 (13.73) | 80.42 (12.55) | 76.72 (15.69)
  Post Infusion - min000 | 81.50 (13.85) | 79.25 (14.77) | 76.22 (16.13)
  Post Infusion - min005 | 77.44 (12.19) | 73.25 (13.97) | 79.06 (16.00)
  Post Infusion - min010 | 77.38 (13.64) | 73.75 (13.60) | 77.78 (15.38)
  Post Infusion - min015 | 75.13 (13.59) | 75.17 (12.71) | 78.83 (14.50)
  Post Infusion - min020 | 78.88 (13.72) | 76.92 (11.24) | 78.39 (14.74)
  Post Infusion - min025 | 79.25 (12.46) | 75.75 (14.14) | 77.44 (12.87)
  Post Infusion - min030 | 80.31 (11.16) | 74.83 (11.76) | 78.33 (13.92)
  Post Infusion - min040 | 80.63 (16.66) | 74.92 (10.42) | 78.39 (13.85)
  Post Infusion - min050 | 79.00 (11.89) | 75.67 (12.20) | 78.33 (14.58)
  Post Infusion - min060 | 78.00 (11.35) | 77.08 (13.21) | 79.11 (13.64)
  Post Infusion - min070 | 78.81 (11.12) | 77.75 (13.92) | 77.50 (13.95)
  Post Infusion - min080 | 80.69 (10.87) | 75.92 (14.85) | 78.06 (14.94)
  Post Infusion - min090 | 80.25 (10.07) | 78.42 (16.55) | 78.89 (14.29)
  Post Infusion - min100 | 80.06 (10.51) | 79.75 (16.80) | 80.17 (14.29)
  Post Infusion - min110 | 79.88 (10.25) | 77.50 (16.94) | 80.22 (14.72)
  Post Infusion - min120 | 80.19 (11.73) | 80.83 (17.02) | 78.44 (14.30)

21. Other Pre Specified Outcome: ECG Measures at All Time Points by Group
Description: Infusion 1 (Day 0) - ECG measures at all time points by group
Time Frame: Day 0 - Baseline (pre-infusion), During Infusion (@30 min), Post-Infusion (@60min)
Population: All subjects receiving a complete or partial Phase 1 infusion
Measure: Mean (Standard Deviation); unit: mm/sec
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 16 | 18
mm/sec
  Baseline_PR Interval | 162.84 (30.09) | 149.11 (11.52) | 164.56 (19.61)
  Baseline_QRS Interval | 91.37 (11.37) | 86.89 (8.76) | 88.11 (10.12)
  Baseline_QT Interval | 380.16 (26.60) | 384.28 (31.47) | 381.94 (36.50)
  Baseline_RR Interval | 0.81 (0.19) | 0.82 (0.15) | 0.81 (0.19)
  30min_PR Interval | 159.63 (34.81) | 152.40 (12.44) | 167.59 (21.30)
  30min_QRS Interval | 89.79 (11.22) | 88.00 (10.39) | 89.12 (9.97)
  30min_QT Interval | 385.11 (25.55) | 385.27 (29.72) | 385.53 (42.92)
  30min_RR Interval | 0.76 (0.12) | 0.81 (0.16) | 0.81 (0.20)
  End_PR Interval | 165.94 (38.63) | 149.43 (11.33) | 165.63 (25.23)
  End_QRS Interval | 91.67 (13.43) | 87.50 (9.63) | 89.00 (10.09)
  End_QT Interval | 371.94 (41.97) | 377.00 (25.33) | 391.13 (43.35)
  End_RR Interval | 0.79 (0.12) | 0.80 (0.11) | 0.82 (0.20)

22. Other Pre Specified Outcome: ECG Measures at All Time Points by Group
Description: Infusion 2 (Day 14) - ECG measures at all time points by group
Time Frame: Day 14 - Baseline (pre-infusion), During Infusion (@30 min), Post-Infusion (@60min)
Population: All subjects receiving a complete or partial Phase 2 infusion
Measure: Mean (Standard Deviation); unit: mm/sec
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 14 | 18
mm/sec
  Baseline_PR Interval | 155.47 (23.46) | 149.46 (15.61) | 167.61 (20.02)
  Baseline_QRS Interval | 92.82 (11.29) | 86.46 (10.05) | 91.33 (12.45)
  Baseline_QT Interval | 379.35 (29.59) | 385.69 (35.84) | 387.33 (38.27)
  Baseline_RR Interval | 0.80 (0.17) | 0.86 (0.16) | 0.84 (0.19)
  30min_PR Interval | 156.18 (21.95) | 146.69 (14.85) | 172.00 (19.76)
  30min_QRS Interval | 90.18 (11.95) | 87.00 (7.98) | 88.44 (10.76)
  30min_QT Interval | 389.18 (25.33) | 360.08 (46.52) | 380.44 (33.30)
  30min_RR Interval | 0.75 (0.11) | 0.77 (0.18) | 0.82 (0.18)
  End_PR Interval | 160.41 (26.48) | 153.55 (19.87) | 165.63 (21.08)
  End_QRS Interval | 95.41 (9.90) | 86.64 (9.90) | 89.50 (9.97)
  End_QT Interval | 387.06 (38.89) | 384.91 (29.89) | 383.25 (31.60)
  End_RR Interval | 0.80 (0.16) | 0.86 (0.11) | 0.81 (0.16)

23. Other Pre Specified Outcome: Incidence of Treatment-Emergent Adverse Events (TEAEs)
Description: Incidence of Treatment-Emergent Adverse Events (TEAE) by Treatment Group. A treatment emergent adverse event (TEAE) is an AE that either began following initiation of study treatment or was present prior to the initiation of the treatment, but increased in frequency or severity following initiation treatment, regardless of causality.
Time Frame: The period of observation for collection of treatment-emergent adverse events extends from Day 0 treatment through the final visit at Day 28.
Population: Number of Treatment-Emergent Adverse Events (TEAEs) in Each Treatment Group
Measure: Number; unit: # of TEAEs
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 16 | 18
# of TEAEs | 13 | 8 | 10

24. Other Pre Specified Outcome: Number of Subject Withdrawals Due to Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 23
Time Frame: The period of observation extends from Day 0 treatment through the final visit at Day 28
Population: All subjects withdrawn from the study due to TEAEs
Measure: Number; unit: participants
Groups:
- Drug - Drug: Phase 1 - intravenous sodium Nitroprusside (SNP) Phase 2 - intravenous sodium Nitroprusside (SNP)
  Subjects will receive i.v. sodium nitroprusside (0.5 μg/kg/min for 4 hours) at Day 0 and Day 14
- Placebo - Drug: Phase 1 - intravenous dextrose (Placebo) Phase 2 - intravenous sodium Nitroprusside (SNP)
  Subjects will receive i.v. placebo (intravenous dextrose) at Day 0 and i.v. sodium nitroprusside (0.5 μg/kg/min for 4 hours) at Day 14
- Placebo - Placebo: Phase 1 - intravenous dextrose (Placebo) Phase 2 - intravenous dextrose (Placebo)
  Subjects will receive i.v. placebo (intravenous dextrose) at Day 0 and again at Day 14.
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 16 | 18
participants | 3 | 4 | 0

25. Other Pre Specified Outcome: Systematic Assessment for Treatment Emergent Effects-Systematic Inquiry (SAFTEE-SI) - Percent of Participants Reporting Experiencing Symptoms at "Moderate" or "Severe" Level for the 10 Most Frequently Reported Symptoms Post Randomization
Description: The Systematic Assessment for Treatment Emergent Effects-Systematic Inquiry (SAFTEE-SI): This is a self-rated 77-item questionnaire organized into 13 body areas assessing possible adverse events during the course of the trial.
Time Frame: Baseline (Day - 1), Follow-Up = reported at any assessment thereafter, including 7 hours after Infusions #1 and #2, Baseline 2 (Day 13) and final follow-up, including early termination visits.
Population: Includes all subjects with SAFTEE data
Measure: Number; unit: percentage of participants
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
Number analyzed (Participants) | 18 | 16 | 18
percentage of participants
  10. Baseline - Hearing or seeing things | 22.2 | 25.0 | 22.2
  10. Follow-Up - Hearing or seeing things | 33.3 | 31.3 | 16.7
  3. Baseline - Feeling drowsy or sleepy | 16.7 | 0.0 | 22.2
  3. Follow-Up - Feeling drowsy or sleepy | 22.2 | 25.0 | 22.2
  8. Baseline - Trouble concentrating | 16.7 | 6.3 | 22.2
  8. Follow-Up - Trouble concentrating | 11.1 | 18.8 | 27.8
  7. Baseline - Poor memory | 11.1 | 6.3 | 27.8
  7. Follow-Up - Poor memory | 5.6 | 25.0 | 22.2
  1. Baseline - Trouble Sleeping | 16.7 | 6.3 | 27.8
  1. Follow-Up - Trouble Sleeping | 11.1 | 12.5 | 22.2
  4. Baseline - Feeling nervous or hyper | 5.6 | 18.8 | 33.3
  4. Follow-Up - Feeling nervous or hyper | 5.6 | 18.8 | 22.2
  18. Baseline - Dry mouth | 5.6 | 12.5 | 11.1
  18. Follow-Up - Dry mouth | 5.6 | 25.0 | 16.7
  34. Baseline - Frequent need to urinate | 0.0 | 6.3 | 11.1
  34. Follow-Up - Frequent need to urinate | 5.6 | 18.8 | 16.7
  17. Baseline - Stuffy nose | 5.6 | 6.3 | 16.7
  17. Follow-Up - Stuffy nose | 5.6 | 18.8 | 11.1
  52. Baseline - Hot flashes | 0.0 | 6.3 | 5.6
  52. Follow-Up - Hot flashes | 11.1 | 6.3 | 16.7

ADVERSE EVENTS:
Time Frame: The period of observation for collection of adverse events extends from the time the subject gave informed consent until the final visit at Day 28.
Arm/Group | Drug - Drug | Placebo - Drug | Placebo - Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 11/23 | 9/19 | 9/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug - Drug (N=23) | Placebo - Drug (N=19) | Placebo - Placebo (N=18)
Hypotension (Cardiac disorders) | 5 | 1 | 1
Headache (Nervous system disorders) | 3 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 2
Chest Pain (Cardiac disorders) | 0 | 1 | 2
Low O2 Saturation Rate (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Abnormal ECG (Cardiac disorders) | 1 | 1 | 0
Decreased Libido (Reproductive system and breast disorders) | 1 | 0 | 1
Dizziness (Vascular disorders) | 0 | 1 | 1
Lightheadedness (General disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 2
Flushing (Vascular disorders) | 2 | 0 | 0
Nausea/Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Increased Appetite (Gastrointestinal disorders) | 1 | 0 | 0
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Drowsiness (General disorders) | 1 | 0 | 0
Dry Mouth (General disorders) | 0 | 0 | 1
Feeling Nervous or Hyperactive (Psychiatric disorders) | 0 | 0 | 1
Hot Flashes (Vascular disorders) | 1 | 0 | 0
Irregular Heart Activity (Cardiac disorders) | 0 | 1 | 0
Pelvic Pain (General disorders) | 0 | 0 | 1
Tingling (Nervous system disorders) | 1 | 0 | 1
White Blood Cell Decrease (Immune system disorders) | 1 | 0 | 0
Blurred Vision (Eye disorders) | 0 | 1 | 0
Elevated ALT Levels (Hepatobiliary disorders) | 0 | 0 | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Heat Exhaustion (General disorders) | 0 | 1 | 0
Hypersomnia (Psychiatric disorders) | 0 | 1 | 0
Increased Heart Rate (Cardiac disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Hypertension (Cardiac disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT02164981/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT02164981/SAP_001.pdf